CLINICAL TRIAL: NCT00239824
Title: Urinary Incontinence After Radical Prostatectomy. - Effect of Pelvic Floor Muscle Training. A Randomised Controlled Trial
Brief Title: Pelvic Floor Muscle Training to Treat Urinary Incontinence After Radical Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Norwegian Fund for Postgraduate Training in Physiotherapy (Other); Fund for Cancer Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REK4.2005.211; T-97450/001
Record Dates: First submitted 2005-10-14; First posted 2005-10-17 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Urinary Incontinence
Keywords: urinary incontinence; pelvic floor muscle training; radical prostatectomy; physiotherapy
MeSH Terms: conditions — Urinary Incontinence | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Strength training of the pelvic floor muscles with follow up instructions by a physiotherapist
  Interventions: Behavioral: Strength training of the pelvic floor muscles; Behavioral: strength training of the pelvic floor muscles with or without follow up instructions by a physiotherapist
- 2 (Active Comparator): Strength training of the pelvic floor muscles without follow up instructions
  Interventions: Behavioral: strength training of the pelvic floor muscles with or without follow up instructions by a physiotherapist

INTERVENTIONS:
Behavioral: Strength training of the pelvic floor muscles — Group A followed a pelvic floor muscle exercise course consisting of intensive pelvic floor muscle training with follow up instructions (training group or DVD instructions)by a physiotherapist;3 x 10 contractions daily.
  Group B were instructed to train the pelvic floor muscles 3 x 10 contractions daily without follow up instructions by a physiotherapist.
  Other Names: Physiotherapy, pelvic floor muscle training
  Arms: 1
Behavioral: strength training of the pelvic floor muscles with or without follow up instructions by a physiotherapist

SUMMARY:
The aim of this study is to evaluate the effect of pelvic floor muscle training in the treatment of urinary incontinence after radical prostatectomy.

DETAILED DESCRIPTION:
Urinary incontinence is a well known side effect of radical prostatectomy. The prevalence differs according to time period after the operation and the definition of incontinence used. However, a prevalence of 10-20% have been reported one year after the operation. Pelvic floor muscle training has been suggested as a treatment of urinary incontinence. The aim of this study is to evaluate the effect of pelvic floor muscle training in the treatment of urinary incontinence after radical prostatectomy.We conduct a randomized clinical trial, comparing one group(n=40) following a pelvic floor muscle training program after prostatectomy and one group (n=40) receiving only standard information.Primary outcome variable is self registration of urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Cancer prostata operated (radical prostatectomy)
* Incontinence after separation of catheter
* Understands Norwegian language

Exclusion Criteria:

* Drug/alcohol abuse

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-10; Primary Completion 2007-12 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
self reported continence (no need for wearing a pad)at 3 months | One year

SECONDARY OUTCOMES:
Self reported time period from operation to continence. | One year
24 hours home pad test registering grams of urine | One year
Pelvic floor muscle strength | one year
Erectile dysfunction | one year
Quality of life | one year
Perceived problems with urinary function | One year

CONTACTS AND LOCATIONS:
Overall Officials: Siv Mørkved, PhD, Study Chair — Clinical Services, St Olavs Hospital/ Dept.of Community Medicine and General Practice, Norwegian University of Science and Technology, Trondheim, Norway
Locations (1):
- Clinical Services, St.Olavs Hospital, Trondheim University Hospital, Trondheim University Hospital, Trondheim, Norway

REFERENCES:
- [Result] Overgard M, Angelsen A, Lydersen S, Morkved S. Does physiotherapist-guided pelvic floor muscle training reduce urinary incontinence after radical prostatectomy? A randomised controlled trial. Eur Urol. 2008 Aug;54(2):438-48. doi: 10.1016/j.eururo.2008.04.021. Epub 2008 Apr 18. PMID 18448233